CLINICAL TRIAL: NCT05369156
Title: The Effects of Chiropractic Care on Neurophysiological Function, Immune Markers and Health-Related Quality of Life in Adults With Subclinical Spinal Pain Using AI Modelling
Brief Title: The Effects of Chiropractic Care in Adults With Subclinical Spinal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REC/01288 Imran Amjad
Record Dates: First submitted 2022-04-26; First posted 2022-05-11 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Subclinical Spinal Pain
Keywords: Subclinical Spinal Pain
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: research
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chiropractic care Group (Experimental): A registered chiropractor will assess the entire spine, and both sacroiliac joints will be assessed for vertebral subluxation by a registered chiropractor with at least five years of clinical experience.The clinical indicators that will be used to assess the function of the spine before spinal adjustment intervention include assessing for joint tenderness to palpation manually palpating for a restricted intersegmental range of motion, assessing for palpable asymmetric intervertebral muscle tension, and any abnormal or blocked joint play and end-feel of the joints. Chiropractors use these biomechanical characteristics as clinical indicators of spinal dysfunction and vertebral subluxation.
  Interventions: Other: Chiropractic Care
- Control Group (Placebo Comparator): The participants head and/or spine will be moved in ways that include passive and active movements, similar to what is done when assessing the spine by a chiropractor. The control intervention will also include the participants moving into adjustment setup positions similar to how the chiropractor would typically set up a patient with no joint pre-loading or adjustive thrust. No spinal adjustment will be performed during any control intervention. This control intervention is not intended to act as a sham treatment session
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Chiropractic Care — The actual force applied to the patient's spine depends on the chiropractor, the patient, and the spinal location of the subluxation, the general shape of the force-time history of spinal adjustments is very consistent and the duration of the thrust is always less than 200 milliseconds.
  Arms: Chiropractic care Group
Other: Control Group — The participants head and/or spine will be moved in ways that include passive and active movements, similar to what is done when assessing the spine by a chiropractor. The sham intervention will also include the participants moving into adjustment setup positions similar to how the chiropractor would typically set up a patient with no joint pre-loading or adjustive thrust
  Arms: Control Group

SUMMARY:
This study aims to investigate long term and retention (in a subgroup) effects of Chiropractic care (CC) on neurological, behavioral, immunological functions and health-related quality of life in adults with subclinical pain.

DETAILED DESCRIPTION:
There is growing evidence that chiropractic care positively impacts various aspects of central and autonomic nervous system function. A single session of chiropractic adjustment has shown to alter pre-frontal cortex (PFC) activity, but there is a lack of robust research investigating the long-term benefits of such PFC changes. This study aims to investigate long term and retention (in a subgroup) effects of Chiropractic care (CC) on neurological, behavioral, immunological functions and health-related quality of life in adults with subclinical pain. In these parallel-group randomized controlled trials, participants aged 18-60 years with subclinical spinal pain will be randomly allocated to receive either 12 weeks of CC intervention or control intervention. Primary outcomes include functional near-infrared spectroscopy, heart rate variability (HRV), serum Brain-Derived Neurotrophic Factors (BDNF) levels and resting-state electroencephalography (EEG). The secondary outcomes include PFC activity (measured by cognitive and behavioral testing), immune and inflammatory markers and health-related quality of life. As data collected in the project is a combination of extrinsic (sociodemographic, clinical questionnaires etc.) and intrinsic physiological data (physiological measures like EEG, HRV etc.), the machine learning or artificial intelligence (AI) will be used to help the development of optimal chiropractic care plans in future.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 60 years
* have subclinical spinal pain

Exclusion Criteria:

* no evidence of spinal dysfunction is present, they are in current pain (above 3/10 on VAS)
* have sought previous treatment for their spinal issues
* are unable to perform the assessment procedures due to contraindications or movement limitations
* diagnosed immune dysfunction
* utilizing a prescribed immunosuppressive medication
* they have uncontrolled asthma
* have nasal polyps
* use of an intranasal steroid spray one month or less before the study
* are HIV-positive
* unable or unwilling to comply with the study protocol
* a history of drug abuse
* are participating in another research study during the time of data collection.
* have any diagnosed comorbidity or concomitant disease
* donated blood within last month
* have allergies to yeast or yeast-derived products
* have chronic sinusitis and/ or recent (within the last six weeks) episodes of acute sinusitis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Functional near-infrared spectroscopy (fNIRS) | Base line
  Functional near-infrared spectroscopy (fNIRS) is an optical imaging tool for noninvasive, continuous monitoring of regional blood flow and tissue oxygenation. It can measure two hemodynamic parameters, both deoxyhemoglobin (HHb) and oxyhemoglobin (HbO2), at the same time. It reflects changes in regional blood flow to areas of the brain involved in processing functional tasks (Cognitive tasks).
  A baseline assessment of a participant will be done before the start of the intervention.
Functional near-infrared spectroscopy (fNIRS) | After 6 weeks
  Functional near-infrared spectroscopy (fNIRS) is an optical imaging tool for noninvasive, continuous monitoring of regional blood flow and tissue oxygenation. It can measure two hemodynamic parameters, both deoxyhemoglobin (HHb) and oxyhemoglobin (HbO2), at the same time. It reflects changes in regional blood flow to areas of the brain involved in processing functional tasks (Cognitive tasks).
  Assessment of participants will be done after 6 weeks of intervention.
Functional near-infrared spectroscopy (fNIRS) | After 12 weeks of intervention
  Functional near-infrared spectroscopy (fNIRS) is an optical imaging tool for noninvasive, continuous monitoring of regional blood flow and tissue oxygenation. It can measure two hemodynamic parameters, both deoxyhemoglobin (HHb) and oxyhemoglobin (HbO2), at the same time. It reflects changes in regional blood flow to areas of the brain involved in processing functional tasks (Cognitive tasks).
  Assessment of participants will be done after 12 weeks of intervention.
Functional near-infrared spectroscopy (fNIRS) | Aftwe 16 weeks of intervention
  Functional near-infrared spectroscopy (fNIRS) is an optical imaging tool for noninvasive, continuous monitoring of regional blood flow and tissue oxygenation. It can measure two hemodynamic parameters, both deoxyhemoglobin (HHb) and oxyhemoglobin (HbO2), at the same time. It reflects changes in regional blood flow to areas of the brain involved in processing functional tasks (Cognitive tasks).
  Assessment of participants will be done after 16 weeks of intervention.
Heart rate variability (HRV) | Up to 16 weeks
  HRV will be used as an objective assessment of psychological health and stress for the participants. High HRV is a marker of an adaptable, responsive nervous system that can detect sensory stimuli and appropriately increase or decrease the heart rate based on the needs of the individual Low HRV and low parasympathetic activity is associated with chronic pain states, poor cardiovascular health and mood disorders.
Serum Brain-derived neurotrophic factor (BDNF) | Base line
  Brain-derived neurotrophic factor (BDNF) plays an important role in neuronal survival and growth, serves as a neurotransmitter modulator, and participates in neuronal plasticity, essential for learning and memory. The higher concentration shows more activity. A baseline assessment of a participant will be done before the start of the intervention.
Serum Brain-derived neurotrophic factor (BDNF) | After 12 weeks of intervention
  Brain-derived neurotrophic factor (BDNF) plays an important role in neuronal survival and growth, serves as a neurotransmitter modulator, and participates in neuronal plasticity, essential for learning and memory. The higher concentration shows more activity. Assessment of participants will be done after 12 weeks of intervention.
Serum Brain-derived neurotrophic factor (BDNF) | After 16 weeks of intervention
  Brain-derived neurotrophic factor (BDNF) plays an important role in neuronal survival and growth, serves as a neurotransmitter modulator, and participates in neuronal plasticity, essential for learning and memory. The higher concentration shows more activity. Assessment of participants will be done after 16 weeks of intervention.
Whole head EEG( sub-cohort of participants) | Base line
  The EEG will be recorded from 40-scalp electrodes using the extended 10-20 system montage (Quick-Cap International). The participant will be seated comfortably in a chair with eyes closed throughout the entire recording. We will record a period of resting whole head EEG. We will use standardized low-resolution brain electromagnetic tomography (sLORETA) for the resting EEG to calculate potential changes (Spatio-spectral Analysis) in brain activity and communication post the chiropractic care intervention. A baseline assessment of a participant will be done before the start of the intervention.
Whole head EEG( sub-cohort of participants) | After 6 weeks of intervention
  The EEG will be recorded from 40-scalp electrodes using the extended 10-20 system montage (Quick-Cap International). The participant will be seated comfortably in a chair with eyes closed throughout the entire recording. We will record a period of resting whole head EEG. We will use standardized low-resolution brain electromagnetic tomography (sLORETA) for the resting EEG to calculate potential changes (Spatio-spectral Analysis) in brain activity and communication post the chiropractic care intervention. Assessment of participants will be done after 6 weeks of intervention.
Whole head EEG( sub-cohort of participants) | After 12 weeks of intervention
  The EEG will be recorded from 40-scalp electrodes using the extended 10-20 system montage (Quick-Cap International). The participant will be seated comfortably in a chair with eyes closed throughout the entire recording. We will record a period of resting whole head EEG. We will use standardized low-resolution brain electromagnetic tomography (sLORETA) for the resting EEG to calculate potential changes (Spatio-spectral Analysis) in brain activity and communication post the chiropractic care intervention. Assessment of participants will be done after 12 weeks of intervention.
Whole head EEG( sub-cohort of participants) | 16 weeks of intervention
  The EEG will be recorded from 40-scalp electrodes using the extended 10-20 system montage (Quick-Cap International). The participant will be seated comfortably in a chair with eyes closed throughout the entire recording. We will record a period of resting whole head EEG. We will use standardized low-resolution brain electromagnetic tomography (sLORETA) for the resting EEG to calculate potential changes (Spatio-spectral Analysis) in brain activity and communication post the chiropractic care intervention.. Assessment of participants will be done after 16 weeks of intervention.

SECONDARY OUTCOMES:
Spatial working memory (SWM) | Base line
  Spatial Working Memory requires retention and manipulation of visuospatial information. This self-ordered test has unique executive function demands and provides a measure of strategy and working memory error.
  Outcome measures include errors (selecting boxes that have already been found to be empty and revisiting boxes that have already been found to contain a token) and strategy. A baseline assessment of a participant will be done before the start of the intervention.
Spatial working memory (SWM) | After 6 weeks of intervention
  Spatial Working Memory requires retention and manipulation of visuospatial information. This self-ordered test has unique executive function demands and provides a measure of strategy and working memory error.
  Outcome measures include errors (selecting boxes that have already been found to be empty and revisiting boxes that have already been found to contain a token) and strategy. Assessment of participants will be done after 6 weeks of intervention.
Spatial working memory (SWM) | After 12 weeks of intervention
  Spatial Working Memory requires retention and manipulation of visuospatial information. This self-ordered test has unique executive function demands and provides a measure of strategy and working memory error.
  Outcome measures include errors (selecting boxes that have already been found to be empty and revisiting boxes that have already been found to contain a token) and strategy. Assessment of participants will be done after 12 weeks of intervention.
Spatial working memory (SWM) | After 16 weeks of intervention
  Spatial Working Memory requires retention and manipulation of visuospatial information. This self-ordered test has unique executive function demands and provides a measure of strategy and working memory error.
  Outcome measures include errors (selecting boxes that have already been found to be empty and revisiting boxes that have already been found to contain a token) and strategy. Assessment of participants will be done after 16 weeks of intervention.
Reaction time (RTI) | Base line
  Reaction Time provides assessments of motor and mental response speeds and measures of movement time, reaction time, response accuracy, and impulsivity.
  Outcome measures are divided into reaction time and movement time for both the simple and five-choice variants.
  More accurate reaction in less time inclines toward good reaction time. A baseline assessment of a participant will be done before the start of the intervention.
Reaction time (RTI) | After 6 weeks
  Reaction Time provides assessments of motor and mental response speeds and measures of movement time, reaction time, response accuracy, and impulsivity.
  Outcome measures are divided into reaction time and movement time for both the simple and five-choice variants.
  More accurate reaction in less time inclines toward good reaction time. Assessment of participants will be done after 6 weeks of intervention.
Reaction time (RTI) | After 12 weeks of intervention
  Reaction Time provides assessments of motor and mental response speeds and measures of movement time, reaction time, response accuracy, and impulsivity.
  Outcome measures are divided into reaction time and movement time for both the simple and five-choice variants.
  More accurate reaction in less time inclines towards good reaction time.Assessment of participants will be done after 12 weeks of intervention.
Reaction time (RTI) | After 16 weeks of intervention
  Reaction Time provides assessments of motor and mental response speeds and measures of movement time, reaction time, response accuracy, and impulsivity.
  Outcome measures are divided into reaction time and movement time for both the simple and five-choice variants.
  More accurate reaction in less time inclines towards good reaction time.Assessment of participants will be done after 16 weeks of intervention.
Paired Associate Learning (PAL) | Base line
  Paired Associates Learning assesses visual memory and new learning. Outcome measures include the errors made by the participant, the number of trials required to locate the pattern(s) correctly, memory scores and stages completed.
  Less errors made by participant shows good memory scores and PAL. A baseline assessment of a participant will be done before the start of the intervention.
Paired Associate Learning (PAL) | After 6 weeks of intervention
  Paired Associates Learning assesses visual memory and new learning. Outcome measures include the errors made by the participant, the number of trials required to locate the pattern(s) correctly, memory scores and stages completed.
  Less errors made by participant shows good memory scores and PAL. Assessment of participants will be done after 6 weeks of intervention.
Paired Associate Learning (PAL) | After 12 weeks of intervention
  Paired Associates Learning assesses visual memory and new learning. Outcome measures include the errors made by the participant, the number of trials required to locate the pattern(s) correctly, memory scores and stages completed.
  Less errors made by participant shows good memory scores and PAL.Assessment of participants will be done after 12 weeks of intervention.
Paired Associate Learning (PAL) | 16 weeks of intervention
  Paired Associates Learning assesses visual memory and new learning. Outcome measures include the errors made by the participant, the number of trials required to locate the pattern(s) correctly, memory scores and stages completed.
  Less errors made by participant shows good memory scores and PAL.Assessment of participants will be done after 16 weeks of intervention.
Stockings of Cambridge (SoC) | Base line
  Stockings of Cambridge (SOC) is a spatial planning test that requires individuals to use problem-solving strategies to match two sets of stimuli Outcome measures include the problem difficulty level reached, mean moves used, and thinking time.
  more of the difficult level reached means participant is more competent and good at problem solving.
Stockings of Cambridge (SoC) | After 6 weeks of intervention
  Stockings of Cambridge (SOC) is a spatial planning test that requires individuals to use problem-solving strategies to match two sets of stimuli Outcome measures include the problem difficulty level reached, mean moves used, and thinking time.
  more of the difficult level reached means participant is more competent and good at problem solving.Assessment of participants will be done after 6 weeks of intervention.
Stockings of Cambridge (SoC) | After 12 weeks of intervention
  Stockings of Cambridge (SOC) is a spatial planning test that requires individuals to use problem-solving strategies to match two sets of stimuli Outcome measures include the problem difficulty level reached, mean moves used, and thinking time.
  more of the difficult level reached means participant is more competent and good at problem-solving.Assessment of participants will be done after 12 weeks of intervention.
Stockings of Cambridge (SoC) | After 16 weeks of intervention
  Stockings of Cambridge (SOC) is a spatial planning test that requires individuals to use problem-solving strategies to match two sets of stimuli Outcome measures include the problem difficulty level reached, mean moves used, and thinking time.
  more of the difficult level reached means participant is more competent and good at problem solving.Assessment of participants will be done after 16 weeks of intervention.
Delayed Matching to Sample (DMS) | Base line.
  Delayed Matching to Sample assesses simultaneous visual matching ability and short-term visual recognition memory for non-verbalizable patterns.
  Outcome measures include latency (the participant's speed of response), the number of correct patterns selected and a statistical measure giving the probability of an error after a correct or incorrect response. A baseline assessment of a participant will be done before the start of the intervention.
Delayed Matching to Sample (DMS) | After 6 weeks of intervention
  Delayed Matching to Sample assesses simultaneous visual matching ability and short-term visual recognition memory for non-verbalizable patterns.
  Outcome measures include latency (the participant's speed of response), the number of correct patterns selected and a statistical measure giving the probability of an error after a correct or incorrect response.Assessment of participants will be done after 6 weeks of intervention.
Delayed Matching to Sample (DMS) | After 12 weeks of intervention
  Delayed Matching to Sample assesses simultaneous visual matching ability and short-term visual recognition memory for non-verbalizable patterns.
  Outcome measures include latency (the participant's speed of response), the number of correct patterns selected and a statistical measure giving the probability of an error after a correct or incorrect response.Assessment of participants will be done after 12 weeks of intervention.
Delayed Matching to Sample (DMS) | After 16 weeks of intervention
  Delayed Matching to Sample assesses simultaneous visual matching ability and short-term visual recognition memory for non-verbalizable patterns.
  Outcome measures include latency (the participant's speed of response), the number of correct patterns selected and a statistical measure giving the probability of an error after a correct or incorrect response. Assessment of participants will be done after 16 weeks of intervention.
Health-Related Quality of life | Baseline
  The health-related quality of life will be measured using the PROMIS-29 v2.0 profile, which assesses pain intensity using a single 0-10 numeric rating item and seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) using four items per domain. The PROMIS-29 v2.0 is a reliable and valid instrument that can be used to assess the impacts of health care interventions and track changes in health over time.
Health-Related Quality of life | After 6 weeks of intervention
  The health-related quality of life will be measured using the PROMIS-29 v2.0 profile, which assesses pain intensity using a single 0-10 numeric rating item and seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) using four items per domain. The PROMIS-29 v2.0 is a reliable and valid instrument that can be used to assess the impacts of health care interventions and track changes in health over time.
Health-Related Quality of life | After 12 weeks of intervention
  The health-related quality of life will be measured using the PROMIS-29 v2.0 profile, which assesses pain intensity using a single 0-10 numeric rating item and seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) using four items per domain. The PROMIS-29 v2.0 is a reliable and valid instrument that can be used to assess the impacts of health care interventions and track changes in health over time.
Health-Related Quality of life | After 16 weeks of intervention
  The health-related quality of life will be measured using the PROMIS-29 v2.0 profile, which assesses pain intensity using a single 0-10 numeric rating item and seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) using four items per domain. The PROMIS-29 v2.0 is a reliable and valid instrument that can be used to assess the impacts of health care interventions and track changes in health over time.

OTHER OUTCOMES:
Immune Function Questionnaire (IFQ) | Base line
  The Immune Function Questionnaire (IFQ) consists of 15 items that assess the frequency of various symptoms associated with poor immune function. There are 19 symptom items included on the questionnaire as signs of weakened immune system functioning: headaches, sore throat, eye infection, sinusitis, runny nose, flu, coughing, cold sores, boils, mild fever, pneumonia, bronchitis, warts/verrucas, sepsis, ear infection, diarrhea, meningitis, sudden high fever, and extended healing injuries. The IFQ score has been found to positively correlate with the number of visits to a General Medical Practitioner. A baseline assessment of a participant will be done before the start of the intervention. Calculate the sum score of the 7 IFQ items. To obtain the final IFQ score, translate the "raw" IFQ scores as follows: Interpretation: 0 = very poor, 10 excellent perceived immune status.
Immune Function Questionnaire (IFQ) | After 6 weeks of intervention
  The IFQ consists of 15 items that assess the frequency of various symptoms associated with poor immune function. There are 19 symptom items included on the questionnaire as signs of weakened immune system functioning: headaches, sore throat, eye infection, sinusitis, runny nose, flu, coughing, cold sores, boils, mild fever, pneumonia, bronchitis, warts/verrucas, sepsis, ear infection, diarrhea, meningitis, sudden high fever, and extended healing injuries. The IFQ score has been found to positively correlate with the number of visits to a General Medical Practitioner. Assessment of participants will be done after 6 weeks of intervention.Calculate the sum score of the 7 IFQ items. To obtain the final IFQ score, translate the "raw" IFQ scores as follows: Interpretation: 0 = very poor, 10 excellent perceived immune status.
Immune Function Questionnaire (IFQ) | After 12 weeks of intervention
  The IFQ consists of 15 items that assess the frequency of various symptoms associated with poor immune function. There are 19 symptom items included on the questionnaire as signs of weakened immune system functioning: headaches, sore throat, eye infection, sinusitis, runny nose, flu, coughing, cold sores, boils, mild fever, pneumonia, bronchitis, warts/verrucas, sepsis, ear infection, diarrhea, meningitis, sudden high fever, and extended healing injuries. The IFQ score has been found to positively correlate with the number of visits to a General Medical Practitioner. Assessment of participants will be done after 12 weeks of intervention. Calculate the sum score of the 7 IFQ items. To obtain the final IFQ score, translate the "raw" IFQ scores as follows: Interpretation: 0 = very poor, 10 excellent perceived immune status.
Immune Function Questionnaire (IFQ) | After 16 weeks of intervention
  The IFQ consists of 15 items that assess the frequency of various symptoms associated with poor immune function. There are 19 symptom items included on the questionnaire as signs of weakened immune system functioning: headaches, sore throat, eye infection, sinusitis, runny nose, flu, coughing, cold sores, boils, mild fever, pneumonia, bronchitis, warts/verrucas, sepsis, ear infection, diarrhea, meningitis, sudden high fever, and extended healing injuries. The IFQ score has been found to positively correlate with the number of visits to a General Medical Practitioner. Assessment of participants will be done after 16 weeks of intervention. Calculate the sum score of the 7 IFQ items. To obtain the final IFQ score, translate the "raw" IFQ scores as follows: Interpretation: 0 = very poor, 10 excellent perceived immune status.
Inflammation markers from Fitbit data | Up to 16 weeks
  Fitbit can be used to measure the autonomic nervous system (ANS). Heart rate variability (HRV) has become a validated marker of autonomic function. In a large population-based study it was found that strong and independent relationships between HR and HRV with a broad set of inflammatory biomarkers. The recording will be done for up to 16 weeks.
Pittsburgh Sleep Quality Index (PSQI) | Base line
  Sleep is also an important determinant of health in general and specifically for stress. PSQI is a reliable self-reported questionnaire to examine the course and natural history of sleep over a 1-month time interval.89 Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as the global score) indicating worse sleep quality.
  A baseline assessment of a participant will be done before the start of the intervention.
Pittsburgh Sleep Quality Index (PSQI) | After 6 weeks of intervention
  Sleep is also an important determinant of health in general and specifically for stress. PSQI is a reliable self-reported questionnaire to examine the course and natural history of sleep over a 1-month time interval.89 Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as the global score) indicating worse sleep quality. Assessment of participants will be done after 6 weeks of intervention.
Pittsburgh Sleep Quality Index (PSQI) | After 12 weeks of intervention
  Sleep is also an important determinant of health in general and specifically for stress. PSQI is a reliable self-reported questionnaire to examine the course and natural history of sleep over a 1-month time interval.89 Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score. Assessment of participants will be done after 12 weeks of intervention. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as the global score) indicating worse sleep quality.
Pittsburgh Sleep Quality Index (PSQI) | After 16 weeks of intervention
  Sleep is also an important determinant of health in general and specifically for stress. PSQI is a reliable self-reported questionnaire to examine the course and natural history of sleep over a 1-month time interval.89 Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as the global score) indicating worse sleep quality.
  Assessment of participants will be done after 16 weeks of intervention.
Depression, Anxiety and Stress Scale -21 (DASS-21) | Base line
  Depression, Anxiety and Stress Scale -21 (DASS-21) is an excellent self-reporting tool for measuring depression, anxiety, and stress features. DASS-21 is a modified version of the full test (DASS-42) with 7 items in each subscale. A baseline assessment of a participant will be done before the start of the intervention. The DASS-21 is the short form of the DASS-42, a self-report scale designed to measure the negative emotional states of depression, anxiety and stress.
Depression, Anxiety and Stress Scale -21 (DASS-21) | After 6 weeks of intervention
  Depression, Anxiety and Stress Scale -21 (DASS-21) is an excellent self-reporting tool for measuring depression, anxiety, and stress features. DASS-21 is a modified version of the full test (DASS-42) with 7 items in each subscale. Assessment of participants will be done after 6 weeks of intervention.
Depression, Anxiety and Stress Scale -21 (DASS-21) | After 12 weeks of intervention
  Depression, Anxiety and Stress Scale -21 (DASS-21) is an excellent self-reporting tool for measuring depression, anxiety, and stress features. DASS-21 is a modified version of the full test (DASS-42) with 7 items in each subscale. Assessment of participants will be done after 12 weeks of intervention.
Depression, Anxiety and Stress Scale -21 (DASS-21) | After 16 weeks of intervention
  Depression, Anxiety and Stress Scale -21 (DASS-21) is an excellent self-reporting tool for measuring depression, anxiety, and stress features. DASS-21 is a modified version of the full test (DASS-42) with 7 items in each subscale. Assessment of participants will be done after 16 weeks of intervention.
International Physical Activity Questionnaire (IPAQ) | Base line
  International Physical Activity Questionnaire (IPAQ) is the most widely used physical activity questionnaire. It measures the duration and frequency of physical activity in the last seven days in different domains. A baseline assessment of a participant will be done before the start of the intervention.
International Physical Activity Questionnaire (IPAQ) | After 6 weeks of intervention
  International Physical Activity Questionnaire (IPAQ) is the most widely used physical activity questionnaire. It measures the duration and frequency of physical activity in the last seven days in different domains. Assessment of participants will be done after 6 weeks of intervention.
International Physical Activity Questionnaire (IPAQ) | After 12 weeks of intervention
  International Physical Activity Questionnaire (IPAQ) is the most widely used physical activity questionnaire. It measures the duration and frequency of physical activity in the last seven days in different domains. Assessment of participants will be done after 12 weeks of intervention.
International Physical Activity Questionnaire (IPAQ) | After 16 weeks of intervention
  International Physical Activity Questionnaire (IPAQ) is the most widely used physical activity questionnaire. It measures the duration and frequency of physical activity in the last seven days in different domains. Assessment of participants will be done after 16 weeks of intervention.
Spine Dysfunction, Stress & Sensory-Motor Integration Questionnaire (SSSMQ) | Base line
  The Spine Dysfunction, Stress & Sensory-Motor Integration Questionnaire is a newly developed tool to assess Spine Dysfunction Characteristics, logical and Psychological Stress Symptoms, and Multimodal and Sensorimotor Integration Dysfunction Symptoms. A higher score on this tool means that respective parameters are on the worse side and lower scores mean respective parameters are on the better side.
  A baseline assessment of a participant will be done before the start of the intervention.
Spine Dysfunction, Stress & Sensory-Motor Integration Questionnaire (SSSMQ) | After 6 weeks of intervention
  The Spine Dysfunction, Stress & Sensory-Motor Integration Questionnaire is a newly developed tool to assess Spine Dysfunction Characteristics, logical and Psychological Stress Symptoms, and Multimodal and Sensorimotor Integration Dysfunction Symptoms. A higher score on this tool means that respective parameters are on the worse side and lower scores mean respective parameters are on the better side. Assessment of participants will be done after 6 weeks of intervention.
Spine Dysfunction, Stress & Sensory-Motor Integration Questionnaire (SSSMQ) | After 12 weeks of intervention
  The Spine Dysfunction, Stress & Sensory-Motor Integration Questionnaire is a newly developed tool to assess Spine Dysfunction Characteristics, logical and Psychological Stress Symptoms, and Multimodal and Sensorimotor Integration Dysfunction Symptoms. A higher score on this tool means that respective parameters are on the worse side and lower scores mean respective parameters are on the better side. Assessment of participants will be done after 12 weeks of intervention.
Spine Dysfunction, Stress & Sensory-Motor Integration Questionnaire (SSSMQ) | After 16 weeks of intervention
  The Spine Dysfunction, Stress & Sensory-Motor Integration Questionnaire is a newly developed tool to assess Spine Dysfunction Characteristics, logical and Psychological Stress Symptoms, and Multimodal and Sensorimotor Integration Dysfunction Symptoms. A higher score on this tool means that respective parameters are on the worse side and lower scores mean respective parameters are on the better side. Assessment of participants will be done after 16 weeks of intervention.
Saliva Cortisol | At baseline
  Salivary cortisol reflects the amount of cortisol that escapes binding proteins and enters the tissues throughout the body, including the salivary glands and saliva.
  For saliva sampling, participants will be requested not to brush their teeth, floss, or eat and drink anything but water for 30 minutes prior to adequate saliva sampling for cortisol assessment.
  Cortisol (otherwise known as the stress hormone) is made in the adrenal glands. It's elevated when we experience heightened anxiety or stress, and it's lowered when we're in a relaxed state. A baseline assessment of a participant will be done before the start of the intervention.
Saliva Cortisol | After 12 weeks of intervention
  Salivary cortisol reflects the amount of cortisol that escapes binding proteins and enters the tissues throughout the body, including the salivary glands and saliva.
  For saliva sampling, participants will be requested not to brush their teeth, floss, or eat and drink anything but water for 30 minutes prior to adequate saliva sampling for cortisol assessment.
  Cortisol (otherwise known as the stress hormone) is made in the adrenal glands. It's elevated when we experience heightened anxiety or stress, and it's lowered when we're in a relaxed state. Assessment of participants will be done after 12 weeks of intervention.
Saliva Cortisol | After 16 weeks of intervention
  Salivary cortisol reflects the amount of cortisol that escapes binding proteins and enters the tissues throughout the body, including the salivary glands and saliva.
  For saliva sampling, participants will be requested not to brush their teeth, floss, or eat and drink anything but water for 30 minutes prior to adequate saliva sampling for cortisol assessment.
  Cortisol (otherwise known as the stress hormone) is made in the adrenal glands. It's elevated when we experience heightened anxiety or stress, and it's lowered when we're in a relaxed state. Assessment of participants will be done after 16 weeks of intervention.
Blood Cortisol | At baseline
  Cortisol is a steroid hormone made by your adrenal glands. It helps your body respond to stress, regulate blood sugar, and fight infections. A blood sample is used to measure cortisol levels.
  The cortisol level may show problems with the adrenal glands or pituitary gland. Cortisol is made by the adrenal glands. A baseline assessment of a participant will be done before the start of the intervention.
Blood Cortisol | After 12 weeks of intervention
  Cortisol is a steroid hormone made by your adrenal glands. It helps your body respond to stress, regulate blood sugar, and fight infections. A blood sample is used to measure cortisol levels.
  The cortisol level may show problems with the adrenal glands or pituitary gland. Cortisol is made by the adrenal glands. Assessment of participants will be done after 12 weeks of intervention.
Blood Cortisol | After 16 weeks of intervention
  Cortisol is a steroid hormone made by your adrenal glands. It helps your body respond to stress, regulate blood sugar, and fight infections. A blood sample is used to measure cortisol levels.
  The cortisol level may show problems with the adrenal glands or pituitary gland. Cortisol is made by the adrenal glands. Assessment of participants will be done after 16 weeks of intervention.
Hair Cortisol | At baseline
  Cortisol is a steroid hormone made by your adrenal glands. It helps your body respond to stress, regulate blood sugar, and fight infections.
  The cortisol level may show problems with the adrenal glands or pituitary gland. Cortisol is made by the adrenal glands. Assessment of participants will be done at the baseline of the study.
Hair Cortisol | After 12 weeks of intervention
  Cortisol is a steroid hormone made by your adrenal glands. It helps your body respond to stress, regulate blood sugar, and fight infections.
  The cortisol level may show problems with the adrenal glands or pituitary gland. Cortisol is made by the adrenal glands. Assessment of participants will be done after 12 weeks of intervention.
Smartphone Gait and Balance Application | Baseline
  The system consists of the following three components: i) a smartphone that has an embedded accelerometer, ii) a belt to house the phone on the lower back, iii) and a smartphone balance application. There are six different tasks that the subject has to perform with the system, like, normal walking up to 6 meters, walking with head movement, standing with eyes open and closed and standing on a compromised surface with eyes open and closed. This app. will calculate mediolateral and anterior-posterior sway during each task. Assessment will be done at baseline.
Smartphone Gait and Balance Application | After 6 weeks
  The system consists of the following three components: i) a smartphone that has an embedded accelerometer, ii) a belt to house the phone on the lower back, iii) and a smartphone balance application. There are six different tasks that the subject has to perform with the system, like, normal walking up to 6 meters, walking with head movement, standing with eyes open and closed and standing on a compromised surface with eyes open and closed. This app. will calculate mediolateral and anterior-posterior sway during each task. Assessment will be done after 6 weeks.
Smartphone Gait and Balance Application | After 12 weeks
  The system consists of the following three components: i) a smartphone that has an embedded accelerometer, ii) a belt to house the phone on the lower back, iii) and a smartphone balance application. There are six different tasks that the subject has to perform with the system, like, normal walking up to 6 meters, walking with head movement, standing with eyes open and closed and standing on a compromised surface with eyes open and closed. This app. will calculate mediolateral and anterior-posterior sway during each task. Assessment will be done after 12 weeks.
Smartphone Gait and Balance Application | After 16 weeks
  The system consists of the following three components: i) a smartphone that has an embedded accelerometer, ii) a belt to house the phone on the lower back, iii) and a smartphone balance application. There are six different tasks that the subject has to perform with the system, like, normal walking up to 6 meters, walking with head movement, standing with eyes open and closed and standing on a compromised surface with eyes open and closed. This app. will calculate mediolateral and anterior-posterior sway during each task.Assessment will be done after 16 weeks.
T-Lymphocytes (CD3) | Baseline
  T-Lymphocytes (CD3) is a protein complex and T cell co-receptor that is involved in activating both the cytotoxic T cell and T helper cells. CD3 are immunoregulatory cells. The concentration of CD3 cells shows the status of the immune system.
T-Lymphocytes (CD3) | After 12 weeks
  T-Lymphocytes (CD3) is a protein complex and T cell co-receptor that is involved in activating both the cytotoxic T cell and T helper cells. CD3 are immunoregulatory cells. The concentration of CD3 cells shows the status of the immune system.
T-Lymphocytes (CD3) | After 16 weeks
  T-Lymphocytes (CD3) is a protein complex and T cell co-receptor that is involved in activating both the cytotoxic T cell and T helper cells. CD3 are immunoregulatory cells. The concentration of CD3 cells shows the status of the immune system.
B-Lymphocytes (CD19) | Baseline
  B-Lymphocytes (CD19) are a biomarker for normal and neoplastic B cells, as well as follicular dendritic cells. CD19 functions as the dominant signalling component of a multimolecular complex on the surface of mature B cells. The concentration of CD19 cells shows the status of the immune system.
B-Lymphocytes (CD19) | After 12 weeks
  B-Lymphocytes (CD19) are a biomarker for normal and neoplastic B cells, as well as follicular dendritic cells. CD19 functions as the dominant signalling component of a multimolecular complex on the surface of mature B cells. The concentration of CD19 cells shows the status of the immune system.
B-Lymphocytes (CD19) | After 16 weeks
  B-Lymphocytes (CD19) are a biomarker for normal and neoplastic B cells, as well as follicular dendritic cells. CD19 functions as the dominant signalling component of a multimolecular complex on the surface of mature B cells. The concentration of CD19 cells shows the status of the immune system.
T-Cell receptor CD4 | Baseline
  CD4 (cluster of differentiation 4) is a glycoprotein that serves as a co-receptor for the T-cell receptor (TCR). CD4 is found on the surface of immune cells such as T helper cells, monocytes, macrophages, and dendritic cells. The expression of CD4 cells shows the status of the immune system.
T-Cell receptor CD4 | After 12 weeks
  CD4 (cluster of differentiation 4) is a glycoprotein that serves as a co-receptor for the T-cell receptor (TCR). CD4 is found on the surface of immune cells such as T helper cells, monocytes, macrophages, and dendritic cells. The expression of CD4 cells shows the status of the immune system.
T-Cell receptor CD4 | After 16 weeks
  CD4 (cluster of differentiation 4) is a glycoprotein that serves as a co-receptor for the T-cell receptor (TCR). CD4 is found on the surface of immune cells such as T helper cells, monocytes, macrophages, and dendritic cells. The expression of CD4 cells shows the status of the immune system.
T-Cell receptor CD8 | Baseline
  CD8 (cluster of differentiation 8) is a transmembrane glycoprotein that serves as a co-receptor for the T-cell receptor (TCR). The CD8 co-receptor plays a role in T cell signalling and aiding with cytotoxic T cell-antigen interactions. The expression of CD8 cells shows the status of the immune system.
T-Cell receptor CD8 | After 12 weeks
  CD8 (cluster of differentiation 8) is a transmembrane glycoprotein that serves as a co-receptor for the T-cell receptor (TCR). The CD8 co-receptor plays a role in T cell signalling and aiding with cytotoxic T cell-antigen interactions. The expression of CD8 cells shows the status of the immune system.
T-Cell receptor CD8 | After 16 weeks
  CD8 (cluster of differentiation 8) is a transmembrane glycoprotein that serves as a co-receptor for the T-cell receptor (TCR). The CD8 co-receptor plays a role in T cell signalling and aiding with cytotoxic T cell-antigen interactions. The expression of CD8 cells shows the status of the immune system.
Interleukin 6 (IL-6) | Baseline
  Interleukin 6 (IL-6) is an interleukin that acts as both a pro-inflammatory cytokine and an anti-inflammatory myokine. The concentration of IL-6 shows the status of the inflammation in the body.
Interleukin 6 (IL-6) | After 12 weeks
  Interleukin 6 (IL-6) is an interleukin that acts as both a pro-inflammatory cytokine and an anti-inflammatory myokine. The concentration of IL-6 shows the status of the inflammation in the body.
Interleukin 6 (IL-6) | After 16 weeks
  Interleukin 6 (IL-6) is an interleukin that acts as both a pro-inflammatory cytokine and an anti-inflammatory myokine. The concentration of IL-6 shows the status of the inflammation in the body.
Tumour Necrosis Factor alpha (TNF alpha) | Baseline
  Tumour Necrosis Factor-alpha (TNF alpha), is an inflammatory cytokine produced by macrophages/monocytes during acute inflammation and is responsible for a diverse range of signalling events within cells, leading to necrosis or apoptosis. The concentration of TNF alpha shows the status of the inflammation in the body.
Tumour Necrosis Factor alpha (TNF alpha) | After 12 weeks
  Tumour Necrosis Factor-alpha (TNF alpha), is an inflammatory cytokine produced by macrophages/monocytes during acute inflammation and is responsible for a diverse range of signalling events within cells, leading to necrosis or apoptosis. The concentration of TNF alpha shows the status of the inflammation in the body.
Tumour Necrosis Factor alpha (TNF alpha) | After 16 weeks
  Tumour Necrosis Factor-alpha (TNF alpha), is an inflammatory cytokine produced by macrophages/monocytes during acute inflammation and is responsible for a diverse range of signalling events within cells, leading to necrosis or apoptosis. The concentration of TNF alpha shows the status of the inflammation in the body.
C-reactive protein (CRP) | Baseline
  C-reactive protein is an annular pentameric protein found in blood plasma, whose circulating concentrations rise in response to inflammation. It is an acute-phase protein of hepatic origin that increases following interleukin-6 secretion by macrophages and T cells.
C-reactive protein (CRP) | After 12 weeks
  C-reactive protein is an annular pentameric protein found in blood plasma, whose circulating concentrations rise in response to inflammation. It is an acute-phase protein of hepatic origin that increases following interleukin-6 secretion by macrophages and T cells.
C-reactive protein (CRP) | After 16 weeks
  C-reactive protein is an annular pentameric protein found in blood plasma, whose circulating concentrations rise in response to inflammation. It is an acute-phase protein of hepatic origin that increases following interleukin-6 secretion by macrophages and T cells.
Interferon-gamma (IFN-γ) | Baseline
  Interferon-gamma (IFN-γ) is a cytokine critical to both innate and adaptive immunity, and functions as the primary activator of macrophages, in addition to stimulating natural killer cells and neutrophils.
Interferon-gamma (IFN-γ) | After 12 weeks
  Interferon-gamma (IFN-γ) is a cytokine critical to both innate and adaptive immunity, and functions as the primary activator of macrophages, in addition to stimulating natural killer cells and neutrophils.
Interferon-gamma (IFN-γ) | After 16 weeks
  Interferon-gamma (IFN-γ) is a cytokine critical to both innate and adaptive immunity, and functions as the primary activator of macrophages, in addition to stimulating natural killer cells and neutrophils.
Natural killer cells (CD56). | Baseline
  CD56 is a fundamental marker in the determination of human natural killer (NK) cell subsets. The degree of CD56 expression is ubiquitously used to define human NK cell maturation, functional, and tissue-specific subsets, yet a unifying implication for the degree of CD56 expression in NK cells remains elusive.
Natural killer cells (CD56). | After 12 weeks
  CD56 is a fundamental marker in the determination of human natural killer (NK) cell subsets. The degree of CD56 expression is ubiquitously used to define human NK cell maturation, functional, and tissue-specific subsets, yet a unifying implication for the degree of CD56 expression in NK cells remains elusive.
Natural killer cells (CD56). | After 16 weeks
  CD56 is a fundamental marker in the determination of human natural killer (NK) cell subsets. The degree of CD56 expression is ubiquitously used to define human NK cell maturation, functional, and tissue-specific subsets, yet a unifying implication for the degree of CD56 expression in NK cells remains elusive.

CONTACTS AND LOCATIONS:
Overall Officials: IMRAN KHAN NIAZI, PhD, Principal Investigator — New Zealand College of Chiropractic
Locations (1):
- Railway General Hospital, Rawalpindi, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Amjad I, Niazi IK, Kumari N, Ghani U, Rashid U, Duarte FCK, Fortuna F, Iglesias S, Gonzalez D, Sumich A, Fabre B, Holt K, Haavik H. The effects of 12 weeks of chiropractic spinal adjustments on physiological biomarkers in adults: A pragmatic randomized controlled trial. PLoS One. 2025 Dec 11;20(12):e0338730. doi: 10.1371/journal.pone.0338730. eCollection 2025. PMID 41379843